CLINICAL TRIAL: NCT05033275
Title: Screening for Sacral Agenesis in Offspring of Mothers With Diabetes in Pregnancy
Status: Terminated | Type: Observational
Why Stopped: Funding ended
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Akshaya Vachharajani, Professor of Pediatrics, University of Missouri-Columbia
Other Study IDs: 2047262
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Infant of Diabetic Mother; Sacral Agenesis
MeSH Terms: conditions — Sacral defect and anterior sacral meningocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Babies born to mothers with pregestational diabetes will be screened with parental consent for sacral agenesis

DETAILED DESCRIPTION:
Parent/s of babies born to mothers with pregestational diabetes who have normal clinical examination and have no radiographs showing a normal sacrum will be approached for a spinal US

ELIGIBILITY:
Inclusion Criteria:

* Infants born to mothers with pregestational diabetes
* Normal spinal examination

Exclusion Criteria:

* Infants born to mothers with pregestational diabetes
* Abnormal spinal examination such as a sacral dimple
* Radiograph with abnormal sacrum
* Spanish speaking parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born to mothers with pregestational diabetes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Babies with sacral agenesis identified with screening of asymptomatic babies with a spinal ultrasound | 12 months
  All babies who have tethered cord on spinal US will be referred to neurosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Akshaya J Vachharajani, MD, Principal Investigator — MU
Locations (1):
- MU, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing

REFERENCES:
- [Derived] Gajagowni S, Mazuru-Witten D, Hegstrom J, Goodman J, Vachharajani AJ. Ultrasound-Guided Prospective Screening for Spinal Dysraphism in Offspring of Mothers With Pregestational Diabetes: A Pilot Study. J Ultrasound Med. 2023 Dec;42(12):2867-2872. doi: 10.1002/jum.16327. Epub 2023 Oct 4. PMID 37792458